CLINICAL TRIAL: NCT00595556
Title: Zonisamide vs. Placebo in the Treatment of Alcohol Dependence
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Albert J. Arias, MD, University of Connecticut Health Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 06-113-1; P50AA003510 (NIH); M01RR006192 (NIH)
Record Dates: First submitted 2008-01-06; First posted 2008-01-16 (Estimated); Results first posted 2010-10-15 (Estimated); Last update posted 2010-10-15 (Estimated); Status verified 2010-09

CONDITIONS: Alcoholism; Alcohol Abuse; Alcohol Dependence
Keywords: Zonisamide; Pharmacotherapy; Alcohol dependence; anticonvulsant
MeSH Terms: conditions — Alcoholism | interventions — Zonisamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Zonisamide
  Interventions: Drug: zonisamide
- B (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: zonisamide — flexible dosages of 100-500mg/day
  Other Names: Zonegran
  Arms: A
Drug: Placebo — Placebo
  Arms: B

SUMMARY:
This is a pilot study designed to examine the potential efficacy and tolerability of zonisamide compared to placebo for the treatment of alcohol dependence.

DETAILED DESCRIPTION:
Zonisamide is an antiepileptic medication which has similar clinical and pharmacologic effects to topiramate, a medication that has demonstrated efficacy in a randomized clinical trial for treatment of alcoholism. Because zonisamide is potentially better tolerated and easier to titrate in the outpatient setting than topiramate, it may offer important clinical advantages in the treatment of alcoholism.

This is a small 12-week placebo-controlled pilot study examining tolerability and potential efficacy in anticipation of a larger, placebo-controlled trial of zonisamide for treatment of alcohol dependence. It is a randomized, double-blind trial of zonisamide vs. placebo at flexible dosages of 100-500mg/day in alcoholics receiving ambulatory psychosocial treatment. Participants will take part in six individual Cognitive-Behavioral based therapy sessions, which are focused on learning coping skills. Participants must endorse a goal of either cutting down their drinking to non-hazardous levels, or abstinence.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 65 years, inclusive
* current Diagnostic & Statistical Manual of Mental Disorders 4th ed (DSM-IV) alcohol dependence (within the past month)
* have 2 heavy drinking days per week during the period between screening and baseline (defined as >4 standard drinks per day for males, and >3 standard drinks per day for females)
* able to read at the eighth grade or higher level and show no evidence of significant cognitive impairment
* if a woman of child-bearing potential (i.e., who has not had a hysterectomy, bilateral oophorectomy, tubal ligation or who is less than two years postmenopausal), must be non-lactating, practicing a reliable method of birth control including barrier method; and have a negative serum pregnancy test prior to initiation of treatment
* be willing to provide signed, informed consent to participate in the study

Exclusion Criteria:

* have a current, clinically significant physical disease or abnormality (i.e., neurologic, renal, rheumatologic, gastrointestinal, hematologic, pulmonary, endocrine, cardiovascular, hepatic, or autoimmune disease that, in the context of the study would represent a risk to the subject, or significant laboratory abnormalities such as hepatic aminotransferase levels greater than 300% of the uper limit of normal or direct bilirubin levels 150% of the upper limit of normal) on the basis of medical history, physician examination, or routine laboratory evaluation. Serum creatinine level of > 1.2 mg/dl will also be exclusionary. Other specific exclusionary disorders include:

  * patients with a history of renal calculi
  * patients with a history of hypersensitivity to zonisamide or any sulfonamide, Stevens-Johnson Syndrome, penicillin allergy, or history of any severe drug allergic reaction
  * patients with a significant history of systemic autoimmune disease such as lupus erythematosis, fibromyalgia, or rheumatoid arthritis
  * patients with a current blood dyscrasia or a history of such, with the exception of a remote history of iron deficient anemia
* have a serious psychiatric illness (i.e., schizophrenia, bipolar disorder, severe or psychotic major depression, panic disorder, or substantial suicide or violence risk) on the basis of history or psychiatric examination
* current dependence on opioids or benzodiazepines or other sedatives will also be exclusionary
* are considered by investigators to be clinically inappropriate for study participation
* because individuals with a history of seizure disorder could potentially be at increased risk of experiencing a seizure due to their drinking, such individuals will also be excluded
* have participated in another pharmacotherapy study in the past thirty days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-07; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Albert J. Arias, MD, Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Zonisamide Medication Treatment: Subjects in this arm received the zonisamide anticonvulsant medication in double blind fashion starting with 100mg daily and titrated every other week to a target dose of 500mg daily. The pills were over-encapsulated to match the placebo.
- Placebo: Subjects in this arm received a double blind placebo lactose capsule identical to the over-capsule on the actual medicine. The titration of "dose" and number of pills matched that of the zonisamide arm.
Period: Overall Study
Arm/Group | Zonisamide Medication Treatment | Placebo
Started | 20 | 20
Completed | 17 | 19
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zonisamide Medication Treatment | Placebo | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 47.8 (9.9) | 50.4 (11) | 49.1 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 12 | 11 | 23
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Change in Number of Heavy Drinking Days (i.e., 5 or More Drinks Per Day for Men, and 4 or More Per Day for Women)Per Week, by Week
Description: This outcome measure represents the change in number of heavy drinking days (i.e., 5 or more drinks per day for men, and 4 or more per day for women)per week, from baseline to the end of week twelve. This was analyzed using weekly measurements over the 12 week study period (thirteen time points, 12 measurements)with a repeated measures analysis (SPSS linear mixed models), by interaction with time (week).
Time Frame: baseline to the end of 12 weeks in treatment
Measure: Mean (Standard Deviation); unit: Days/week
Arm/Group | Zonisamide Medication Treatment | Placebo
Number analyzed (Participants) | 20 | 20
Days/week | -.30 (.362) | -.20 (.362)
Statistical Analysis 1: Comparison: Zonisamide Medication Treatment vs Placebo; Test type: Superiority or Other; p = .012, Mixed Models Analysis

2. Primary Outcome: Weekly Rate of Change in Abstinent Days
Description: This outcome measure analyzed the weekly rate of change in number of abstinent days over the twelve weeks of the study from baseline to the end of week twelve. This was analyzed using weekly measurements over the 12 week study period (thirteen time points, 12 measurements)with a repeated measures analysis (SPSS proc mixed), by interaction with time (week).
Time Frame: baseline to the end of 12 weeks in treatment
Measure: Mean (Standard Error); unit: days/week
Arm/Group | Zonisamide Medication Treatment | Placebo
Number analyzed (Participants) | 20 | 20
days/week | 0.17 (.02) | 0.13 (.02)
Statistical Analysis 1: Comparison: Zonisamide Medication Treatment vs Placebo; Test type: Superiority or Other; p = .94, Mixed Models Analysis

3. Secondary Outcome: Change in Number of Drinks Per Week by Week
Description: This outcome measure represents the change in the total number of standard drinks per week (weekly data) from baseline to the end of week twelve. This was analyzed using weekly measurements from baseline to week 12 week of the study period (thirteen time points, 12 measurements)with a repeated measures analysis (SPSS linear mixed models), by interaction with time (week).
Time Frame: baseline to the end of 12 weeks in treatment
Population: The analysis was intention to treat and last observation carried forward
Measure: Mean (Standard Deviation); unit: drinks/week
Arm/Group | Zonisamide Medication Treatment | Placebo
Number analyzed (Participants) | 20 | 20
drinks/week | -2.2 (20.5) | -1.4 (20.5)
Statistical Analysis 1: Comparison: Zonisamide Medication Treatment vs Placebo; Test type: Superiority or Other; p = .004, Mixed Models Analysis

4. Secondary Outcome: Change in the Urge to Drink Alcohol as Measured by the Alcohol Urge Questionnaire (AUQ)
Description: This is the change in measured urge to drink alcohol as measured by the Alcohol Urge Questionnaire (AUQ), measured every 2 weeks from baseline until the last week of the study (over twelve weeks, 7 timepoint measurements of AUQ, 6 calculated changes). It is reported in terms of change per visit (every 2 weeks). AUQ measures a feeling state, and uses a 7 point (1-7)Likert scale for each of 8 items (questions). The lowest urge score is 8 (representing less urge to drink), and the highest would be tabulated as 56 (meaning more urge to drink). Repeated measures SPPS linear mixed models used.
Time Frame: baseline to the end of 12 weeks in treatment
Measure: Mean (Standard Deviation); unit: units on a scale/visit
Arm/Group | Zonisamide Medication Treatment | Placebo
Number analyzed (Participants) | 20 | 20
units on a scale/visit | -1.4 (1) | -0.6 (1)
Statistical Analysis 1: Comparison: Zonisamide Medication Treatment vs Placebo; Test type: Superiority or Other; p = .006, Mixed Models Analysis

5. Secondary Outcome: Change in Gamma-glutamyl Transferase (GGT) Concentration
Description: This outcome measure looks at the change in blood levels of this enzyme assay from baseline, and then after 6 weeks (midpoint), and then at the endpoint (12 weeks). The analysis takes into account all three time points, and reports the average change between each of the three time points.
Time Frame: 12 weeks (from initiation to end of treatment)
Measure: Mean (Standard Deviation); unit: Units/Liter
Arm/Group | Zonisamide Medication Treatment | Placebo
Number analyzed (Participants) | 20 | 20
Units/Liter | 8.4 (36.2) | 2.9 (36.2)
Statistical Analysis 1: Comparison: Zonisamide Medication Treatment vs Placebo; Test type: Superiority or Other; p = .3, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 14 weeks
Arm/Group | Zonisamide Medication Treatment | Placebo
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 16/20 | 16/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zonisamide Medication Treatment (N=20) | Placebo (N=20)
GI (Gastrointestinal disorders) | 13 (16) | 4 (5)
Neurologic (Nervous system disorders) | 8 (10) | 5 (5)
Psychiatric (Psychiatric disorders) | 4 (4) | 8 (14)
Cognitive (Nervous system disorders) | 4 (4) | 2 (2)
Genitourinary (Reproductive system and breast disorders) | 4 (4) | 2 (2)
Fatigue/Somnolence (General disorders) | 4 (6) | 1 (1)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)

LIMITATIONS AND CAVEATS:
The small sample size and the short duration of treatment are limitations. High rates of retention in the treatment and adherence to the medication regimen are strengths. The concomitant psychotherapy may have caused a ceiling effect on medication.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No